CLINICAL TRIAL: NCT05082870
Title: Using a Psychosocial Transitional Group to Improve Adaptation, Coping and Mental Health Outcomes Following Limb Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1517
Record Dates: First submitted 2021-09-16; First posted 2021-10-19 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Amputation
Keywords: Group Intervention; Limb Loss; Feasibility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Research Coordinator and Statistician analyzing the data will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive-expressive group therapy (Experimental): The SEGT approach fosters mutual support, promotes openness and emotional expression. SEGT will be delivered and co-facilitated by a psychiatrist and an allied healthcare professional. It is a 6-module program held over a 3-week period (approximately 2 hour sessions X 2 week) that is framed within social cognitive theory, whereby resilience to adversity (limb loss in this instance) relies on personal enablement.
  Interventions: Behavioral: Supportive-expressive group therapy (SEGT)
- Treatment as usual (No Intervention): The treatment as usual group will receive standard care only (which may include an individual psychiatric consultation).

INTERVENTIONS:
Behavioral: Supportive-expressive group therapy (SEGT) — The SEGT approach fosters mutual support, promotes openness and emotional expression. SEGT will be delivered and co-facilitated by a psychiatrist and an allied healthcare professional. It is a 6-module program held over a 3-week period (approximately 2 hour sessions X 2 week) that is framed within social cognitive theory, whereby resilience to adversity (limb loss in this instance) relies on personal enablement.
  Arms: Supportive-expressive group therapy

SUMMARY:
People with limb loss receiving inpatient rehabilitation are at greater risk for depression and anxiety, social isolation, and generally have poor quality of life. To proactively address the mental health needs of this population, this study plans to test an innovative psychological group therapy program designed for limb loss inpatients to enhance coping skills, address mental health challenges, and better prepare them to integrate back into the community via a randomized blinded feasibility trial. Since this is a novel intervention, adapted specifically for limb loss, this study will test the feasibility of delivering this inpatient group program to these at-risk individuals to see: if they will participate in the program, what they like/do not like about it, and if there are some early findings suggesting it is effective. Researchers will use these results to improve the psychosocial group program and to further test its effectiveness in a larger clinical study.

DETAILED DESCRIPTION:
Lower limb extremity amputation (LEA) is a debilitating event that negatively affects many aspects of an individual's life, such as their mobility, physical and mental health, and ultimately quality of life (QoL). Due to the high rates of diabetes in Canada, the most common type of limb loss is dysvascular due to complications of diabetes/vascular disease.

Compared to other limb loss populations (trauma or tumor), people with dysvascular LEA have been shown to have poorer QoL. Premorbid comorbidities (e.g. coronary heart disease, etc.), and post-morbid complications such as depression, anxiety and chronic pain further impact wellbeing. Sequelae of these issues include impaired body image, and high rates of suicidal ideation. Rates of depression have been found to be as high as 60%; comorbid depression is associated with lower prosthetic use, higher perceived vulnerability, and lower self-rated overall health. Providers, however, often focus efforts on the patients' physical recovery post-LEA and may not adequately address psychosocial functioning.

There is some preliminary evidence on the efficacy of group therapy approaches for limb loss patients undergoing inpatient rehabilitation in India, and outpatient rehabilitation in Canada, but findings are limited and may not be fully generalizable to dysvascular LEA.

Hence, the planned innovative intervention will provide clarification on the feasibility of undertaking a larger scale trial to assess the efficacy of an inpatient group therapy approach to address the mental health concerns (i.e., depression and anxiety) and psychosocial needs (i.e. coping skills) of limb loss patients. Based on available knowledge, this would be the first of its kind in Canada.

ELIGIBILITY:
Patient Inclusion Criteria:

* English-speaking adult inpatients (18 years and older)
* Dysvascular-related lower extremity amputation
* Medically stable
* No clinical suspicion of cognitive impairment
* No history of active psychosis or unstable severe mental health diagnosis (no diagnosis of schizophrenia, dementia, etc.)
* Admitted inpatients to St. John's Rehab Hospital (Sunnybrook Health Sciences Centre).

Patient Exclusion Criteria:

* Actively suicidal
* Unable participate effectively in a group setting
* Non-dysvascular lower extremity amputation
* Non-English-speaking
* Children (under the age of 18)
* Medically unstable
* Clinical suspicion of cognitive impairment
* History of active psychosis or unstable severe mental health diagnosis (diagnosis of schizophrenia, dementia, etc.)

Staff Inclusion Criteria: (Note: Staff will not be part of intervention, but will be asked to share their perspectives on the intervention)

* Clinical staff who work on the inpatient A1 unit at St. John's Rehab (Sunnybrook Health Sciences Centre)

Staff Exclusion Criteria:

* Casual or contract staff who have worked on the inpatient A1 unit.
* Non-St. John's Rehab Hospital staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Participant recruitment | Through study completion, an average of 1 year.
  Number of participants who are recruited into the study and are contacted for assessments at set time intervals.
Questionnaire completion rates | At 3 months post-discharge for SEGT and control group.
  Number of completed assessments.
Treatment adherence | Through study completion, an average of 1 year.
  Number of participants who complete all 6 SEGT sessions.
Number of participants contacted for follow up interview | At 1 month-post discharge for SEGT group
  Number of participants contacted for follow up interview
Participant retention | At three months post-discharge for SEGT and control group
  Number of participants who complete the 3 month post-discharge assessments
Participant retention | At one month post-discharge for SEGT group
  Number of participants who complete 1 month post-discharge interview

SECONDARY OUTCOMES:
Change in Depression and Anxiety | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Hospital Anxiety and Depression Scale: The HADS is a 14-item depression and anxiety screening tool that asks participants to rank the severity of their depression and anxiety symptoms using a 4-point scale (0 to 3). Scores are summed for anxiety items (HADS-A) and for the depression items (HADS-D) with higher scores indicating greater severity of symptoms. The scores are interpreted as normal (range: 0-7), borderline abnormal (range: 8-10), and abnormal (range: 11-21).
Change in Self-efficacy | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Coping Self-Efficacy Scale:The CSES is a measures perceived self-efficacy for coping with challenges and threats. It is a 26-item measure rated using an 11-point scale with the anchors 0 (cannot do at), 5 (moderately certain can do), and 10 (certain can do). Total scores are calculated by summing the item scores and a higher score indicates higher coping self-efficacy.
Change in Body image | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Amputee Body Image Scale-Revised: The ABIS-R is a measure of body image perception in people living with limb loss. The measure consists of 14-items scored using the scale 0 (none of the time), 1 (sometimes), and 2 (most/all of the time). Total scores are obtained by reverse scoring three items and summing the item scores.
Change in Health-related quality of life | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  Short Form-36 Survey: The SF-36 is the most widely used generic health-related QoL tool. The tool measures 8 domains including physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, social functioning, general mental health, role limitations due to emotional problems, and vitality. Higher scores on the measure are indicative of less disability.
Change in Community participation | A. 3 months post-discharge
  Reintegration to Normal Living Index: The RNLI assesses involvement in recreational and social activities, perceived ability to move within the community, and the degree of comfort people have with their relationships. The measure consists of 11 statements and participants are asked to rate each statement on a scale from 1 (Does not describe my situation) to 10 (Fully describes my situation). An adjusted score is calculated producing a score range of 0-100.
Psychiatric consultations | Through study completion, an average of 1 year.
  # of individual psychiatric consultations

CONTACTS AND LOCATIONS:
Overall Officials: Rosalie Steinberg, MSC, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pezzin LE, Dillingham TR, MacKenzie EJ. Rehabilitation and the long-term outcomes of persons with trauma-related amputations. Arch Phys Med Rehabil. 2000 Mar;81(3):292-300. doi: 10.1016/s0003-9993(00)90074-1. PMID 10724073
- [Background] Fortington LV, Dijkstra PU, Bosmans JC, Post WJ, Geertzen JH. Change in health-related quality of life in the first 18 months after lower limb amputation: a prospective, longitudinal study. J Rehabil Med. 2013 Jun;45(6):587-94. doi: 10.2340/16501977-1146. PMID 23624575
- [Background] Turner AP, Meites TM, Williams RM, Henderson AW, Norvell DC, Hakimi KN, Czerniecki JM. Suicidal ideation among individuals with dysvascular lower extremity amputation. Arch Phys Med Rehabil. 2015 Aug;96(8):1404-10. doi: 10.1016/j.apmr.2015.04.001. Epub 2015 Apr 14. PMID 25883037
- [Background] Amtmann D, Morgan SJ, Kim J, Hafner BJ. Health-related profiles of people with lower limb loss. Arch Phys Med Rehabil. 2015 Aug;96(8):1474-83. doi: 10.1016/j.apmr.2015.03.024. Epub 2015 Apr 25. PMID 25917819
- [Background] Bilandzic A, Rosella L. The cost of diabetes in Canada over 10 years: applying attributable health care costs to a diabetes incidence prediction model. Health Promot Chronic Dis Prev Can. 2017 Feb;37(2):49-53. doi: 10.24095/hpcdp.37.2.03. PMID 28273040
- [Background] Moxey PW, Gogalniceanu P, Hinchliffe RJ, Loftus IM, Jones KJ, Thompson MM, Holt PJ. Lower extremity amputations--a review of global variability in incidence. Diabet Med. 2011 Oct;28(10):1144-53. doi: 10.1111/j.1464-5491.2011.03279.x. PMID 21388445
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Padovani MT, Martins MR, Venancio A, Forni JE. Anxiety, depression and quality of life in individuals with phantom limb pain. Acta Ortop Bras. 2015 Mar-Apr;23(2):107-10. doi: 10.1590/1413-78522015230200990. PMID 27069411
- [Background] McDonald S, Sharpe L, Blaszczynski A. The psychosocial impact associated with diabetes-related amputation. Diabet Med. 2014 Nov;31(11):1424-30. doi: 10.1111/dme.12474. Epub 2014 May 24. PMID 24766143
- [Background] Fleury AM, Salih SA, Peel NM. Rehabilitation of the older vascular amputee: a review of the literature. Geriatr Gerontol Int. 2013 Apr;13(2):264-73. doi: 10.1111/ggi.12016. Epub 2012 Dec 26. PMID 23279009
- [Background] Horgan O, MacLachlan M. Psychosocial adjustment to lower-limb amputation: a review. Disabil Rehabil. 2004 Jul 22-Aug 5;26(14-15):837-50. doi: 10.1080/09638280410001708869. PMID 15497913
- [Background] Schaffalitzky E, Gallagher P, Maclachlan M, Ryall N. Understanding the benefits of prosthetic prescription: exploring the experiences of practitioners and lower limb prosthetic users. Disabil Rehabil. 2011;33(15-16):1314-23. doi: 10.3109/09638288.2010.529234. Epub 2010 Nov 4. PMID 21050130
- [Background] Srivastava K, Chaudhury S. Rehabilitation after amputation: psychotherapeutic intervention module in Indian scenario. ScientificWorldJournal. 2014 Jan 12;2014:469385. doi: 10.1155/2014/469385. eCollection 2014. PMID 24526895
- [Background] Delehanty RD, Trachsel L. Effects of short-term group treatment on rehabilitation outcome of adults with amputations. International Journal of Rehabilitation and Health. 1995;1(2):61-73.